CLINICAL TRIAL: NCT05660044
Title: Human Factors Validation Study of Artificial Intelligence Ultrasound Navigation Software for Cardiac Imaging
Brief Title: Human Factors Study of Ultrasound Navigation Software for Cardiac Imaging
Status: Completed | Type: Observational
Sponsor: UltraSight (Industry)
Responsible Party: Sponsor
Other Study IDs: USEG 301
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-06

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Product is a machine learning software, that utilizes AI to provide real-time guidance to acquire diagnostic-quality ultrasound views of the heart.

DETAILED DESCRIPTION:
Participants are healthcare professionals, who are not performing echocardiography on a routine basis. Participants attend a short training session to learn the software, then have a memory-decay period, followed by an individual simulated-use scanning session, lasting up to 60 minutes with a Moderator at the heart institute.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Novice users or medical professionals who do not perform echocardiographs as part of their routine job responsibilities.
* Have the capacity to understand study risks and consent to be in the study
* Be available and willing to participate in the study
* Not be employed by the Sponsor or another medical device or pharmaceutical company

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 28-34 study participants will be recruited to meet at least one of the following professions:
  * Attending Physicians and/or Medical Residents
  * Registered Nurses (RNs), Nurse Practitioners (NPs) and Physician Assistants (PAs)
  * Medical assistants (CMAs)
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Usability of UltraSight AI guidance software | 10 days
  Demonstrate that the Product can be used by the intended users by a questionnaire that is filled by an observation moderator which will assess the ease of use and user satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Danny Spiegelstein, MD, Study Director — UltraSight
Locations (1):
- Sheba medical center, Ramat Gan, Israel